CLINICAL TRIAL: NCT06131320
Title: Visuo-spatial Profile in Children with Cerebral Palsy Born At Term or Not and Anatomical Correlation
Brief Title: Brain Lesion and Visuospatial Impairment in CP Child
Acronym: EVSP-ANAT-CP
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1053
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Children with Cerebral Palsy
Keywords: Cerebral Palsy, child, visuo-spatial disorder, brain lesion
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CP child
  Interventions: Diagnostic Test: PVSE Test; Other: Cerebral MRI
- CP child with a PVSE test and a cerebral MRI performed during his/her follow-up
  Interventions: Diagnostic Test: PVSE Test; Other: Cerebral MRI

INTERVENTIONS:
Diagnostic Test: PVSE Test — Completion of the PVSE test
Other: Cerebral MRI — Cerebral MRI scan

SUMMARY:
Children with cerebral palsy (CP) show varying degrees of motor impairment and movement disorders whose perceptive-visual contribution has yet to be established. The literature reports that children with CP have more frequent neuro-visual disorders. The link between the location and size of the brain lesion and neurovisual symptomatology has yet to be explored.

In this retrospective clinical data study, we will investigate in children with PC whether there is an anatomo-clinical correlation between visuo-spatial disorders is the brain injury of interest to the dorsal visual pathway. We will explore the volume of grey and white matter parietal involvement.

To test visuo-spatial disorders, we will use the PVSE (Visuo-Spatial Elementary Perception) test which does not require motor skills or language and is therefore suitable for children with a PC. This test will make it possible to better identify the deficit or deficits in order to adapt an early remediation. It could serve as a reference for comparing several pathologies/etiologies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 4 to 18 yo
* With a CP diagnosis
* With PVSE test completion during his/her regular follow-up
* With a cerebral MRI scan during his/her regular follow-up

Exclusion Criteria:

- With an incomplete PVSE test or whose interpretation was deemed unreliable by the rater

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children coming for out-patient consultation at the paediatric rehabilitation unit of the Hospices Civils de Lyon for a CP diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
PVSE test results: total score and 8 sub-scores (length perception, size perception, angle comparison, midline localization, position perception, position selection, occipital score and parietal score.) | At the inclusion
  Using normative values of PVSE test, we assess pathological measure inferior outlier limits and subnormal measure below the lower quartile limit

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric rehabilitation unit of the Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No